CLINICAL TRIAL: NCT01266434
Title: The Additive Anti-inflammatory Effect of Simvastatin in Combination With Inhaled Corticosteroids on p38 MAPK in Asthma
Acronym: Simvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Kittipong Maneechotesuwan, Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: si481/2010
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Asthma
Keywords: moderate persistent asthma; Inhaled corticosteroids
MeSH Terms: conditions — Asthma | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- simvastatin (Experimental)
  Interventions: Drug: Simvastatin
- B1-6-12 (Placebo Comparator)
  Interventions: Drug: Simvastatin; Drug: B1-6-12

INTERVENTIONS:
Drug: Simvastatin — 10 mg once daily for 8 weeks
  Other Names: Zocor
Drug: B1-6-12 — 1 tablet once daily for 8 weeks
  Arms: B1-6-12

SUMMARY:
To test whether simvastatin has an additional anti-inflammatory effects on p38 MAPK, a signaling molecule for inflammation in inhaled steroid-treated asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* mild-to-moderate persistent asthmatics
* FEV1 = OR > 50% of predicted

Exclusion Criteria:

* Previous history of renal disease or serum creatinine is more than 2 mg/dl.
* Previous history of liver disease.
* Pregnancy or lactation.
* Are already receiving or are known to be allergic to statins or to have developed myositis.
* Have an asthma exacerbation requiring treatment with oral corticosteroids during the 3 months prior to the commencement of study entry.
* Being treated with immunosuppressive agents.
* Unwilling to cooperate the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Sputum eosinophils | 8 weeks
  To determine the additive effect of simvastatin on airway inflammation in ICS-treated patients with persistent asthma by measuring eosinophil counts in induced sputum and on lung function (FEV1)

SECONDARY OUTCOMES:
Phosphorylated p38 MAPK in sputum cells | 8 weeks
  1. To determine the additional effects of simvastatin in combination with inhaled corticosteroids on the expression of phosphorylated p38 MAPK and phosphorylated activating transcription factor (ATF)2 in induced sputum cells from asthmatic patients.
  2. To confirm the above in vivo results in the in vitro model using monocyte-derived dendritic cells.
  3. To determine the effects of simvastatin and/or corticosteroids on Th2 cytokine production by peripheral blood CD4+ T-lymphocytes in vitro.

CONTACTS AND LOCATIONS:
Overall Officials: Kittipong - Maneechotesuwan, MD., PhD., Principal Investigator — Siriraj Hospital
Locations (1):
- Division of Respiratory Disease and TB, Siriraj Hospital, Bangkoknoi, BKK, Thailand